CLINICAL TRIAL: NCT01362543
Title: Treatment With Cognitive Behavioural Therapy in Traumatised Refugees - Stress Management Versus Cognitive Restructuring - a Randomised Clinical Trial
Brief Title: Traumatized Refugees -Stress Management Versus Cognitive Re-structuring
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mental Health Centre Copenhagen, Bispebjerg and Frederiksberg Hospital (Other)
Collaborators: University of Copenhagen (Other)
Responsible Party: Principal Investigator, Jessica Carlsson Lohmann, M.D., Phd, Mental Health Centre Copenhagen, Bispebjerg and Frederiksberg Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PTF2
Record Dates: First submitted 2011-05-24; First posted 2011-05-30 (Estimated); Last update posted 2014-05-14 (Estimated); Status verified 2014-05

CONDITIONS: Posttraumatic Stress Disorder
Keywords: PTSD; Depression; Refugees; Trauma
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Depression; Wounds and Injuries | interventions — Cognitive Behavioral Therapy; Cognitive Restructuring

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Stress Management (Active Comparator)
  Interventions: Other: Cognitive behavioural therapy (stress management)
- Cognitive restructuring (Active Comparator)
  Interventions: Other: Cognitive Behavioural Therapy (cognitive restructuring)

INTERVENTIONS:
Other: Cognitive behavioural therapy (stress management) — Following a manual
  Arms: Stress Management
Other: Cognitive Behavioural Therapy (cognitive restructuring) — Following a manual
  Arms: Cognitive restructuring

SUMMARY:
The Competence Centre for Transcultural Psychiatry is a clinic specialised in the treatment of traumatised refugees. There is a lack of studies on treatment effect in traumatised refugees. There are several studies indicating an effect of cognitive behavioural therapy (CBT) in Posttraumatic Stress Disorder (PTSD). A few studies point to that CBT could be effective in traumatised refugees. There are no studies examining if some methods used in CBT are more useful than others in traumatised refugees. The aim of this study is to examine the effect of CBT with focus on Stress Management versus cognitive restructuring. Patients included in this study will be randomised to either Stress Management or cognitive restructuring. All referred patients will receive medical treatment as usual (described in the clinic's manual for medical doctors, 2011). All patients that fulfill the inclusion criteria will be included in the study. Hopefully this study will contribute to improve the psychotherapeutic treatment offered to traumatised refugees.

ELIGIBILITY:
Inclusion Criteria:

* Refugee or patient that has been reunified with family member being a refugee.
* Symptoms of PTSD in accordance with International Classification of Diseases-10 (ICD-10) research criteria.
* Trauma in the past such as imprisonment, torture (according to UN definition), war experiences.
* Referred by a medical doctor.
* Motivated for treatment.
* Informed consent.

Exclusion Criteria:

* Severe psychotic illness such as schizophrenia or bipolar disorder
* Drug abuse
* Patients admitted to in ward treatment
* No informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 143 (Actual)
Dates: Start 2011-06; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Change in PTSD symptoms measured by the first 16 items in the Harvard Trauma Questionnaire (HTQ) | Baseline, after 2 months and after 6 months

SECONDARY OUTCOMES:
Change in depressive symptoms measured by the Hopkins Symptoms Checklist-25 (HSCL-25), depressive items | Baseline, after 2 months and after 6 months
Change in anxiety symptoms measured by the Hopkins Symptom Checklist-25 (HSCL-25), anxiety items | Baseline, after 2 months and after 6 months
Change in quality of life measured by the WHO-5 | Baseline, after 2 months and 6 months
Changes in functioning measured by the the Sheehan Disability Scale (SDS) | Baseline, after 2 months and 6 months
Achievement of goals set at beginning of psychotherapy using Goal Attainment Scaling (GAS) | After 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Jessica M Carlsson Lohmann, MD, PhD, Principal Investigator — Competence Centre for Transcultural Psychiatry
Locations (1):
- Competence Centre for Transcultural Psychiatry, Ballerup Municipality, Denmark

REFERENCES:
- See also: Link to web page of the Competence Centre for Transcultural Psychiatry (mostly in Danish) — http://www.psykiatri-regionh.dk/menu/Centre/Psykiatriske+centre/Psykiatrisk+Center+Ballerup/Undersogelse+og+behandling/Kompetencecenter+for+Transkulturel+Psykiatri/